CLINICAL TRIAL: NCT03856034
Title: In Utero Endoscopic Correction of Myelomeningocele: Laparotomy Versus Percutaneous - A Pilot Study
Brief Title: Laparotomy Versus Percutaneous Endoscopic Correction of Myelomeningocele
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: USFetus (Other)
Collaborators: Wellington Hospital (Other Government); University of Southern California (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1249628
Record Dates: First submitted 2019-02-05; First posted 2019-02-27 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Neural Tube Defects; Spina Bifida; Myelomeningocele; Chiari Malformation
Keywords: spina bifida; myelomeningocele; neural tube defect; chiari malformation; fetoscopy; percutaneous; fetus
MeSH Terms: conditions — Neural Tube Defects; Spinal Dysraphism; Meningomyelocele; Arnold-Chiari Malformation | interventions — Fetoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Fetoscopic repair (Experimental)
  Interventions: Device: Fetoscopy

INTERVENTIONS:
Device: Fetoscopy — Patients will receive fetoscopic repair of myelomeningocele. Patients with an anterior placenta will undergo the laparotomy with uterine exteriorization approach. Patients with a posterior placenta will undergo the percutaneous approach (or, if patient prefers, the laparotomy with uterine exteriorization approach).

SUMMARY:
The purpose of this study is to evaluate the feasibility of a fetoscopic surgical technique for antenatal correction of fetal myelomeningocele. Two surgical approaches will be utilized. The percutaneous approach will be offered to participants with a posterior placenta. The laparotomy/uterine exteriorization approach will be offered to participants regardless of placental location.

ELIGIBILITY:
Inclusion Criteria:

1. Myelomeningocele (including myeloschisis) at level T1 through S1 with hindbrain herniation. Lesion level and hindbrain herniation will be confirmed by MRI and ultrasonography.
2. Maternal age ≥18 years.
3. Gestational age of 19 to 27 6/7 weeks' gestation as determined by clinical information and evaluation of first ultrasound.
4. Balanced karyotype with written confirmation of culture results. Results by fluorescence in situ hybridization (FISH) will be acceptable if the patient is at 24 weeks or more.
5. Positive evaluation of social work consult indicating the patient is capable of consenting to the procedure and has the appropriate social support system to participate in the study.
6. Positive evaluation from pediatric neurology consult.
7. Willing to remain in the greater Wellington or Pasadena area (within a 30-minute car ride) for remainder of the pregnancy and deliver at Wellington Regional Medical Center or Huntington Memorial Hospital for postnatal management. The participants must be willing to return to our center for the 12, 24, 30, 48, and 60 months for follow-up evaluation.

Exclusion Criteria:

1. Multiple gestation
2. Insulin-dependent pregestational diabetes
3. Presence of a fetal anomaly not related to myelomeningocele. A fetal echocardiogram will be conducted before surgery and if the finding is abnormal, the patient will be excluded.
4. Fetal kyphosis of 30 degrees or more, assessed by ultrasound or MRI.
5. Presence of uterine cervical cerclage or history of incompetent cervix.
6. Placenta previa or placental abruption.
7. Short cervix < 25 mm measured by cervical ultrasound.
8. Obesity as defined by body mass index (BMI) of 35 or greater.
9. History of previous spontaneous singleton delivery prior to 37 weeks.
10. Maternal-fetal Rh isoimmunization, Kell sensitization or a history of neonatal alloimmune thrombocytopenia.
11. Maternal HIV or Hepatitis-B status positive because of the increased risk of transmission to the fetus during maternal-fetal surgery. If the patient's HIV or Hepatitis B status is unknown, the patient must be tested and found to have negative results before she can be enrolled.
12. Known Hepatitis-C positivity. If the patient's Hepatitis C status is unknown, she does not need to be screened.
13. Uterine anomaly such as large (greater than 6 cm) fibroids, cervical fibroids or multiple fibroids or Mullerian duct abnormality.
14. Other maternal medical condition which is a contraindication to surgery or anesthesia.
15. Patient does not have a support person (e.g., husband, partner, parents).
16. Inability to comply with the travel and follow-up requirements of the study.
17. Patient does not meet psychosocial criteria as determined by the social worker evaluation.
18. Participation in another intervention study that influences maternal and fetal morbidity and mortality.
19. Maternal hypertension as determined by the investigator, which would increase the risk of preeclampsia or preterm delivery (including, but not limited to: uncontrolled hypertension, chronic hypertension with end organ damage and new onset hypertension in current pregnancy).
20. Bicornuate uterus or any other uterine malformation the PI decides is not safe for surgery.
21. Nickel allergy.
22. Maternal request to undergo open fetal surgery for the antenatal correction of open spina bifida at our institution primarily or after failed fetoscopic approach.
23. Known maternal hypersensitivity to bovine collagen or chondroitin materials.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2018-11-02 (Actual); Primary Completion 2020-11-02 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of successful in-utero fetoscopic myelomeningocele closures using either laparotomy or percutaneous techniques | At time of surgery until delivery, up to 21 weeks
  Successful fetoscopic closure of the spinal defect and reversal of hindbrain herniation as assessed by ultrasound and MRI prior to delivery

CONTACTS AND LOCATIONS:
Overall Officials: Ruben Quintero, MD, Principal Investigator — Wellington Regional Medical Center; Ramen Chmait, MD, Principal Investigator — University of Southern California/ Huntington Memorial Hospital
Locations (2):
- United States (2):
  - University of Southern California / Huntington Memorial Hospital, Los Angeles, California
  - Wellington Regional Medical Center, Wellington, Florida

IPD SHARING:
Plan to Share IPD: No